CLINICAL TRIAL: NCT03877458
Title: Combined Probiotics is More Effective in the Treatment of Infantile Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shu-Fen Wu, Attending physician, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMUH105-REC1-155
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Infantile Colic
Keywords: Infantile Colic; Bifidobacteria and Lactobacilli; Intestinal Microbiome; Probiotics
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- L. acidophilus TYCA06, B. longum BLI-02 and B. bifidum VDD088 (Experimental): Taking 1 mix probiotics capsule at bed time everyday for three months.
  Interventions: Other: L. acidophilus TYCA06, B. longum BLI-02 and B. bifidum VDD088
- L. reuteri GL-104 (Experimental): Taking 1 probiotic capsule at bed time everyday for three months.
  Interventions: Other: L. reuteri GL-104
- Placebo group (Placebo Comparator): Taking 1 Placebo capsule at bed time everyday for three months.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: L. acidophilus TYCA06, B. longum BLI-02 and B. bifidum VDD088 — Taking 1 mix probiotics capsule at bed time everyday for three months.
  Arms: L. acidophilus TYCA06, B. longum BLI-02 and B. bifidum VDD088
Other: L. reuteri GL-104 — Taking 1 probiotic capsule at bed time everyday for three months.
  Arms: L. reuteri GL-104
Other: Placebo — Taking 1 placebo capsule at bed time everyday for three months.
  Arms: Placebo group

SUMMARY:
All participants are randomized into 1 of 3 treatment arms, the mixture L acidophilus, B longum and B. bifidum group, Lactobacillus reuteri or placebo group.

Primary outcome is defined as a reduction in the duration of average crying and fussing times, from baseline (day 0) to age 6 months, to <3 hours per day. Secondary outcome are the number of participants who respond to treatment on days 7, 14, 21, 28 and each month till age 6 months.

DETAILED DESCRIPTION:
Infantile colic or excessive infant crying with no medical cause is a burdensome condition. Although crying is often considered "normal behavior," 5%-40% of infants cry inconsolably and excessively, accompanied by bouts of fussiness and gas passing.

The etiology of infantile colic remains unclear; various theories have been proposed, however, recent studies have implicated a potential role of the intestinal microbiome ,colicky infants presents lower amounts of Bifidobacteria and Lactobacilli. Several randomized clinical trials (RCT) have been conducted to examine the effectiveness of Lactobacillus reuteri DSM17938 vs placebo in the treatment of infantile colic. However, there is no trial adopt probiotics contained Bifidobacteria and Lactobacilli to treat infantile colic. In view of the above evidences, the investigators thus hypothesis that probiotics contained Bifidobacteria and Lactobacilli will more effect to increase the diversity of intestinal microbiome and alleviate infantile colic. The objective of this study is to evaluate the efficacy of combine probiotics (L. acidophilus, B. longus and B. bifidus) compare to Lactobacillus reuteri in the treatment infantile colic. Fecal calprotectin levels and microbial community in colic infants before and after probiotics will be evaluated to explore the mechanism of effectiveness of probiotics.

This, double-blind RCT will be carried out from December 2016 to November 2018 at Children's hospital of China Medical university. Eligible infants are included in the study after written informed consent is obtained from a parent/guardian. Study participants will meet the following inclusion criteria: (1) diagnosis of infantile colic (ie, crying or fussy/gassy episodes ≥3 hours/day for ≥3 days/7 days, as defined by a modified definition of Wessel criteria) at study commencement; (2) age 3 weeks to 5 months at study commencement (although infantile colic typically manifests between age 2 weeks and 3-4 months, to capture infants with delayed onset of colic, infants with colic up to 6 months were eligible); (3) exclusively breastfed; (4) term delivery (≥37 weeks gestation); and (5) healthy infants with birth weight ≥2500 g. Exclusion criteria included: (1) a major medical problem or acute illness, including gastroesophageal reflux, as determined by a pediatrician; (2) history of antibiotic treatment before or during the study; (3) history of probiotic supplementation; (4) history of any allergies to any of the ingredients in the probiotic mixture of acidophilus, B longus and B. bifidus or placebo (sunflower oil, medium-chain triglyceride oil, and silicon dioxide); and (5) concurrent participation in another clinical trial.

Primary outcome is defined as a reduction in the duration of average crying and fussing times, from baseline (day 0) to age 6 months, to <3 hours per day. Secondary outcome are the number of participants who respond to treatment on days 7, 14, 21, 28 and each month till age 6months.

All participants are randomized into 1 of 3 treatment arms, the mixture L acidophilus, B longus and B. bifidus group, Lactobacillus reuteri or placebo group. Independent Research Support Pharmacy personnel, not participating in the study at the pharmacy of the Children Hospital prepare a computer-generated 3-treatment randomization schedule with a random block of varying size to ensure balance in the allocation of participants between treatment arms. Stool bacterial microbiota will be accessed by next generation sequence and fecal calprotectin will be measured by ELISA.

A minimum of 60 participants per study arm is needed to provide 80% power to detect an effect size of 0.5 and a detectable difference between groups in mean crying and fussing times of 50 minutes. Statistical analyses are performed using SPSS version 20 (IBM, Armonk, New York) using an intention-to-treat approach. The Student t test is used to compare mean values of continuous variables approximating a normal distribution, and the Mann-Whitney U test is used for nonnormally distributed variables. Proportions are compared using the χ2 test or Fisher exact test, as appropriate. All reported statistical tests are 2-sided.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of infantile colic (ie, crying or fussy/gassy episodes ≥3 hours/day for ≥3 days/7 days, as defined by a modified definition of Wessel criteria) at study commencement.
2. Age 3 weeks to 3 months at study commencement.
3. Infants are born in full term (greater than 37 weeks) and the birth weight more than 2500 grams.

Exclusion Criteria:

1. A major medical problem or acute illness, including gastroesophageal reflux, as determined by a pediatrician.
2. History of antibiotic treatment before or during the study.
3. History of probiotic supplementation.
4. History of any allergies to any of the ingredients in the probiotic mixture of L. acidophilus, B. longum and B. bifidum or placebo.
5. Concurrent participation in another clinical trial.

Ages: 3 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Average crying and fussing times. | 6 months.
  Change in the duration of average crying and fussing times from baseline (day 0) to age 6 months, to <3 hours per day.

SECONDARY OUTCOMES:
The number of participants. | 6 months.
  The number of participants who respond to treatment on days 7, 14, 21, 28 and each month till age 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-chih Lin, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan